CLINICAL TRIAL: NCT07237750
Title: iWAIST Trial: A Multicenter, Open Label, Randomized Controlled Trial Evaluating the Efficacy and Safety of Endoscopic Radial Compression Gastroplasty (ERCG) Versus Optimized Lifestyle Intervention for Weight Loss in Chinese Adults With Overweight or Obesity
Brief Title: iWAIST Trial: ERCG (Endoscopic Radial Compression Gastroplasty) vs Optimized Lifestyle Intervention for Weight Loss
Acronym: iWAIST-RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Liu Yan (Other)
Collaborators: Wuhan TongJi Hospital (Other); The Second Affiliated Hospital of Zhejiang Chinese Medical University (Other); Ankang City Central Hospital (Other); The First Affiliated Hospital of Soochow University (Other); First Affiliated Hospital of Lanzhou University (Unknown)
Responsible Party: Sponsor-Investigator, Liu Yan, Principal Investigator, Department of Gastroenterology, Chinese PLA General Hospital, Beijing 302 Hospital
Organization: Beijing 302 Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 307-2026-iWAIST-RCT
Record Dates: First submitted 2025-09-16; First posted 2025-11-20 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Overweight and/or Obesity; Metabolic Syndrome; Nonalcoholic Fatty Liver Disease; Chinese
Keywords: Endoscopic gastroplasty; Endoscopic bariatric therapy; Weight loss; Overweight; Gastric volume reduction; Chinese; Obesity
MeSH Terms: conditions — Metabolic Syndrome; Non-alcoholic Fatty Liver Disease; Weight Loss; Overweight; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERCG + OLI (Experimental): Sutureless endoscopic gastric volume reduction using a clip-and-loop apposition system under general anesthesia or deep sedation, plus standardized OLI (dietary counseling, calorie deficit, physical activity prescription, and behavioral support) with visit frequency matched to the comparator.
  Interventions: Procedure: Endoscopic Radial Compression Gastroplasty; Behavioral: Optimized Lifestyle Intervention (OLI)
- OLI (Active Comparator): Structured lifestyle program including individualized nutrition counseling targeting a 【~500-750 kcal/day】 deficit, physical activity prescription (≥150 min/week moderate-intensity plus resistance training twice weekly), and behavioral support delivered at the same schedule as the experimental arm.
  Interventions: Behavioral: Optimized Lifestyle Intervention (OLI)

INTERVENTIONS:
Procedure: Endoscopic Radial Compression Gastroplasty — Sutureless endoscopic gastric volume reduction using a novel clip-and-endoloop apposition system; performed under general anesthesia or deep sedation; standard perioperative care.
  Arms: ERCG + OLI
Behavioral: Optimized Lifestyle Intervention (OLI) — Structured nutrition counseling, calorie deficit plan, physical activity prescription per regional guidelines, and behavioral support; visit frequency matched to the ERCG arm.

SUMMARY:
Obesity and overweight are rising in Chinese populations, where metabolic risks begin at lower BMI thresholds than in Western cohorts. Many individuals with overweight or mild-to-moderate obesity are ineligible or unwilling to undergo bariatric surgery due to invasiveness and risk. Endoscopic bariatric and metabolic therapies offer minimally invasive alternatives but vary in complexity, cost, and safety profiles. Investigators developed a sutureless endoscopic procedure, Endoscopic Radial Compression Gastroplasty (ERCG), which reduces gastric volume by apposing gastric walls using a clip-and-loop system. This randomized controlled trial evaluates the efficacy and safety of ERCG versus an optimized lifestyle intervention in Asian adults with BMI 24.0-37.4 kg/m² who have not succeeded with conservative measures. Preliminary studies suggest ERCG can achieve approximately 12% total body weight loss (TBWL) at 3 months. The primary endpoint is percent TBWL at 3 months; secondary outcomes include changes in BMI, metabolic parameters, quality of life, and adverse events. Results are expected to inform the role of ERCG as a safe, effective, and scalable option between conservative care and bariatric surgery.

DETAILED DESCRIPTION:
The prevalence of obesity and overweight continues to increase worldwide, and Chinese populations are particularly vulnerable due to lower thresholds for metabolic risk compared with Western populations. Individuals with overweight or mild-to-moderate obesity (BMI 24.0-37.4 kg/m²) often fail conservative measures but are ineligible or unwilling to undergo bariatric surgery because of its invasiveness, risk, and costs. This creates an unmet need for minimally invasive, effective, and scalable interventions.

Endoscopic bariatric and metabolic therapies (EBMTs) have emerged as alternatives, but many existing procedures involve technically complex endoscopic suturing, high costs, or device-related risks. Investigators developed ERCG, a novel endoscopic procedure that reduces gastric volume by apposing the gastric walls using a newly designed clip-and-loop system. Preliminary studies demonstrated that ERCG can induce rapid weight loss, with mean percent total body weight loss (TBWL) of approximately 12% at 3 months, while maintaining a favorable safety profile.

This randomized controlled trial aims to evaluate the efficacy and safety of ERCG compared with an optimized lifestyle intervention (OLI) in Chinese adults with overweight and mild-to-moderate obesity who have failed conservative weight reduction efforts. Eligible participants will be randomized 1:1 into two groups. The experimental group will undergo ERCG under general anesthesia or deep sedation, following a standardized perioperative protocol, then receive structured OLI. The control group will receive structured OLI consisting of individualized dietary counseling, caloric restriction, exercise prescription, and behavioral support. Follow-up visits are scheduled at 1 month, 2 month, 3 month and 6 month after enrollment.

The primary endpoint is percent TBWL at 3 months, assessed using standardized weight measurement protocols. Secondary endpoints include %EBWL at 3 and 6 months, changes in BMI, metabolic parameters (fasting plasma glucose, HbA1c, insulin resistance indices, lipid profile), quality of life assessed by validated questionnaires (IWQOL-Lite), and the incidence of adverse events classified according to international standards.

Randomization will be computer-generated with concealed allocation, and outcome assessors will be blinded to treatment assignment. Analyses will follow the intention-to-treat principle with appropriate methods for handling missing data.

The study is expected to generate high-quality evidence regarding the short-term and medium-term efficacy of ERCG, to clarify its safety profile, and to determine whether ERCG can serve as a safe and scalable option bridging the therapeutic gap between conservative lifestyle approaches and bariatric surgery for overweight and mildly to moderately obese Chinese populations.

ELIGIBILITY:
Inclusion Criteria:

* Asian adults aged 18-65 years.
* BMI 24.0-37.4kg/m²(Chinese standard)。
* Failed prior conservative weight loss attempts ≥2 months。
* Willingness to comply with follow-up.
* Provided written informed consent.

Exclusion Criteria:

* Prior gastrointestinal surgery with clinically relevant sequelae.
* Active or clinically significant gastrointestinal disease, including inflammatory conditions (e.g., esophagitis, Barrett's esophagus, Crohn's disease), peptic ulcer disease (gastric/duodenal ulcer), or neoplastic lesions.
* Any condition associated with an increased risk of upper gastrointestinal bleeding.
* Hiatal hernia >2 cm or severe/refractory gastroesophageal reflux disease (GERD); acid reflux requiring ≥2 medications for symptom control.
* Esophageal/pharyngeal structural abnormalities that may impede endoscope passage (e.g., stricture, diverticulum).
* Achalasia or other severe esophageal motility disorder.
* Severe coagulopathy.
* Insulin-dependent diabetes mellitus.
* Chronic abdominal pain.
* Gastrointestinal motility disorder (e.g., gastroparesis).
* Hepatic impairment or cirrhosis.
* Severe or uncontrolled psychiatric illness.
* Alcohol abuse or substance dependence.
* Unwilling to participate in a physician-supervised diet/behavior modification program and/or unwilling to comply with routine follow-up.
* Daily regular use of NSAIDs, anticoagulants, or other gastric-irritating medications.
* Unable or unwilling to take proton pump inhibitor (PPI) therapy as prescribed during the treatment period.
* Known or suspected hypersensitivity to any material/component of the study system.
* Pregnant or breastfeeding.
* Severe cardiopulmonary disease or other serious systemic/organic disease.
* Positive Helicobacter pylori (H. pylori) test.
* Use of time-critical medications potentially affected by altered gastric emptying (e.g., antiepileptics, antiarrhythmics).
* Current systemic corticosteroids, immunosuppressants, or opioid analgesics.
* Use of any weight-loss medication within the past 3 months or current use.
* Prior use of any intragastric device.
* Participation in a weight-affecting clinical trial within the past 6 months.
* Symptomatic congestive heart failure, clinically significant arrhythmia, or unstable coronary artery disease.
* Clinically significant respiratory disease.
* Autoimmune connective tissue disease.
* Life expectancy <1 year or severe renal/hepatic/pulmonary or other serious medical illness.
* Known genetic or endocrine cause of obesity (e.g., hypothyroidism, Prader-Willi syndrome) or other endocrine disease known to affect body weight.
* Eating disorder (e.g., night eating syndrome, bulimia nervosa, binge eating disorder, compulsive eating).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Percent Total Body Weight Loss (%TBWL) | 1-6 months post-intervention
  %TBWL = [(Baseline weight - Follow-up weight) / Baseline weight] × 100. Measured using calibrated scale under standardized conditions.
Clinical Responder Rate (CRR) | 3 month, 6 month
  Percentage of participants with %TBWL > 5% at 3/6 months, where %TBWL = [(baseline weight - month 3/6 weight) / baseline weight] × 100.

SECONDARY OUTCOMES:
Body Weight (kg) | Baseline, 1 month, 2 month, 3 month, 6month
  Weight measured on a calibrated scale under standardized conditions (light clothing, no shoes, preferably morning after ≥8h fasting).
Body Height (m) | Baseline
  Standing height measured with a wall-mounted stadiometer, no shoes, heels together, Frankfurt plane horizontal.
Percent Excess Body Weight Loss (%EBWL) | 1-6 months post-intervention
  %EBWL is calculated as [(Baseline weight - Follow-up weight) / (Baseline weight - Ideal weight)] × 100. Ideal weight is defined as the weight corresponding to a BMI of 23.9 kg/m². Weight is measured using a calibrated scale under standardized fasting conditions at each visit.
Change in BMI (kg/m²) | Baseling, 1 month, 2 months, 3 months and 6 months
  BMI will be calculated as weight (kg) divided by height squared (m²).
Glycated Hemoglobin (HbA1c) | Baseline, 3 months
  HbA1c will be measured using standard laboratory methods. Values at each visit and changes from baseline will be summarized.
Adverse Events (AEs/SAEs) Related to Procedure | 3, 6, 12 months
  Number and proportion of participants with device-/procedure-related AEs/SAEs, graded by Clavien-Dindo and per FDA/ISO definitions.
GERD-Q Total Score | Baseline, 3, and 6 months
  Gastroesophageal Reflux Disease Questionnaire (GERD-Q) total score, validated 6-item instrument. Higher scores indicate more severe reflux symptoms.
Postoperative Pain (VAS/NRS) | 6 hours, 24 hours, and 7 days
  Patient-reported pain intensity using a 0-10 scale (0=no pain, 10=worst imaginable pain). Assessed at rest.
Postoperative Nausea Score | 6 hours, 24 hours, and 7 days
  Patient-reported nausea severity using a 0-10 numeric rating scale (0=no nausea, 10=worst nausea).
Total Cholesterol | Baseline, 3 months
  Total cholesterol will be measured after an overnight fast using standard laboratory methods. Values at each visit and changes from baseline will be summarized.
Low-Density Lipoprotein Cholesterol (LDL-C) | Baseline, 3 months
  LDL-C will be measured directly or calculated using standard methods. Values at each visit and changes from baseline will be summarized.

CONTACTS AND LOCATIONS:
Locations (1):
- The fifth Medical Center of Chinese PLA General Hospital, Beijing, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided